CLINICAL TRIAL: NCT05993975
Title: Effects of Intrathecal Dexmedetomidine as an Adjuvant to Low Dose Hyperbaric 0.5% Bupivacaine on Hemodynamic Parameters in Patients Undergoing Transurethral Resection of the Prostate
Brief Title: Effects of Intrathecal Dexmedetomidine as an Adjuvant to Low Dose Hyperbaric 0.5% Bupivacaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sindh Institute of Urology and Transplantation (Other)
Responsible Party: Principal Investigator, Syed Muhammad Abbas, Associate Professor, Department of Anaesthesia, Sindh Institute of Urology and Transplantation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SAbbas
Record Dates: First submitted 2023-07-01; First posted 2023-08-16 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Group BUPPURE will receive 1.5 ml of hyperbaric 0.5% bupivacaine (1.5 ml/7.5 mg) whereas the BUPIDEX group will receive Dexmedetomidine 3 micrograms (0.3mL)with hyperbaric 0.5% bupivacaine (1.2 ml/6 mg) to be given to one group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BUPIPURE (Active Comparator): Hyperbaric Bupivacaine 0.5% (1.5 ml/7.5 mg) to be given intrathecally
  Total volume 1.5 mL
  Interventions: Drug: Bupivacain 0.5%
- BUPI-DEX (Experimental): Hyperbaric Bupivacaine 0.5% (1.2 ml/6 mg)+Dexmedetomidine (0.3 mL) 3 microgram intrathecally.
  Total volume 1.5 mL
  Interventions: Drug: Bupivacain 0.5%; Drug: Dexmedetomidine Hydrochloride

INTERVENTIONS:
Drug: Bupivacain 0.5% — Bupivacaine hydrochloride was given without any adjuvant
  Other Names: Pure Bupivacain 0.5%
Drug: Dexmedetomidine Hydrochloride — Use of Dexmedetomidine Hydrochloride 5 micrograms (1 mL) as an adjuvant with bupivacaine hydrochloride
  Other Names: Dexmedetomidine 5 microgram
  Arms: BUPI-DEX

SUMMARY:
Patients will be enrolled in one of the two groups using a computer-generated random number table: Group I will receive 1.5 ml of 0.5% hyperbaric bupivacaine (7.5 mg). Group II will receive 1.2 mL of 0.5% hyperbaric bupivacaine (6 mg) along with 0.3 mL (3 μg )of dexmedetomidine (total 1.5 mL).

DETAILED DESCRIPTION:
After approval of the synopsis and permission from the hospital ethics committee, all patients meeting the inclusion criteria will be included in the study. Patients will be instructed not to consume solid food after midnight before surgery and to take clear liquids up to 2 hours before surgery. Using a computer-generated random number table, patients will be enrolled in one of the two groups: Group I will receive 1.5 ml of 0.5% hyperbaric bupivacaine (7.5 mg). Group II will receive 1.2 mL of 0.5% hyperbaric bupivacaine (6 mg) along with 0.3 mL (5 μg )of dexmedetomidine (total of 1.5 mL). They will be randomly allocated into two groups using the sealed envelope technique by a person blinded to the procedure. The study medication will be prepared by an anaesthesiologist not involved in the study and another anaesthesiologist performing the spinal block will record the intraoperative and postoperative data. On arrival at the Operating Room (OR) monitors like a non-invasive blood pressure monitor (NIBP), peripheral oxygen saturation monitor (SpO2), and electrocardiography monitor (ECG) having lead II will be attached. All the baseline values of blood pressure (SBP, DBP, and MAP), heart rate and rhythm, and SPO2 will be observed and recorded. An intravenous (IV) line will be established with an 18-gauge cannula. The study drug solutions will look identical. For Group I, 7.5 mg(1.5 mL) of 0.5% hyperbaric bupivacaine hydrochloride will be drawn in a 3 mL BD syringe. For Group II, 6mg (1.3 mL) of 0.5% hyperbaric bupivacaine hydrochloride will be drawn in a 3 mL BD syringe. By using an insulin syringe, 0.3 mL (3 μg) of Dexmedetomidine (preservative free) 100 μg/mL will be added to the 6 mg (1.3 mL) of hyperbaric bupivacaine under complete aseptic conditions to bring the total volume to 1.5 mL. The total volume of drug solutions will be 1.5 mL in each group.

Local infiltration of the skin with 2mL of 2% lidocaine will be done to decrease the discomfort caused by the spinal needle. A spinal puncture will be performed at L3-L4 or L4-L5 with a midline approach using a 25-gauge Quincke needle in the sitting position. After verification of clear and free flow of cerebrospinal fluid, the drug will be administered and the patients will be placed in the supine position Vitals will be monitored Heart Rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), respiratory rate (RR), oxygen saturation (SpO2) for every 5 minutes till the end of surgery. If mean arterial pressure (MAP) decreases below 65 mmHg or the Heart rate falls below 65 beats per minute then intravenous vasopressors will be given. The sensory block levels will be checked on the bilateral mid-clavicular line with a pin prick with a blunt needle every 2 min from the time of drug injection until the sensory level achieves up to T10 level.

In contrast, the motor block will be assessed using the modified Bromage scale. The surgeon will be asked to start the surgery when the sensory block has reached the T10 level. After completion of the surgery, the patient will be shifted to the PACU and monitored for 3 hours with continuous ECG monitoring and intermittent non-invasive blood pressure monitoring at 5-minute intervals. All untoward events like shivering, nausea vomiting, sedation, and respiratory depression will be monitored and recorded in the operating room as well as in the recovery room.

All data will be recorded on Performa attached as Annex A after the consultant anesthetist confirms.

ELIGIBILITY:
Inclusion Criteria:

* ASA I to ASA II
* Age 50 to 80 years old
* Height between 155cm and 175 cm

Exclusion Criteria:

* History of spine surgery or the presence of an infectious focus on the back
* Patient's refusal to undergo a spinal anaesthesia
* Hypersensitivity to bupivacaine or dexmedetomidine
* Patients taking drugs of abuse or narcotic analgesics
* Diabetic neuropathy
* History of bleeding disorders
* Oral/intravenous anticoagulant therapy
* History of arrhythmias or labile hypertension
* Unco-operative patients
* Hearing defect
* ASA III and IV
* Central or peripheral nervous system disorders
* Severe hypovolemia

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients coming for transurethral resection of the prostate
Enrollment: 108 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Height of sensory block | 0 to 4 hours
  Dermatome level having absence of cold sensation
Motor block | 0 to 4 hours
  According to Bromage scores
  Grade Criteria I Free movement of legs and feet II Just able to flex knees with free movement of feet III Unable to flex knees, but with free movement of feet IV Unable to move legs or feet
  we need paralysis of both legs (Bromage score IV) for surgery
Time for 2 segment regression of sensory block | 0 to 4 hours
  Dermatome level having absence of cold sensation
Heart rate | 0 to 4 hours
  By anaesthesia ECG monitor
Mean Blood pressure | 0 to 4 hours
  Non invasive blood pressure monitoring devise

SECONDARY OUTCOMES:
Shivering | 0 to 4 hours
  Bedside Shivering Assessment Score (BSAS) grade 0, if there is no shivering grade 1 if there is no muscle contraction but mild fasciculation of face or neck or peripheral vasoconstriction but no visible shivering, grade 2 if there is a visible muscular activity in only one muscle group, grade 3 if the muscular activity is in more than one muscle group but not generalized grade 4 if gross muscular activity involving the entire body.
  Grade 0 is better, increase in grade (0 -> 4) means worsening

CONTACTS AND LOCATIONS:
Overall Officials: Ali A Lanewala, MD, PhD, Study Director — Sindh Institute of Urology & Transplantation
Locations (1):
- Syed Muhammad Abbas, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No